CLINICAL TRIAL: NCT04080700
Title: Korean Prospective Registry for Evaluating the Safety and Efficacy of Distal Radial Approach (KODRA)
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Seung Hwan Lee, Professor, Wonju Severance Christian Hospital
Other Study IDs: KODRA
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Radial Artery; Puncture
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distal radial approach — Operator puncture the distal radial artery with open needle or venipuncture catheter needle for coronary angiography and percutaneous coronary intervention.

SUMMARY:
The left distal radial approach (DRA) has been introduced as a feasible and safe alternative route of the radial artery. However, there is still lack of evidence for DRA regarding the feasibility, safety, effective time for hemostasis and hemostasis method. This prospective multicenter registry aimed to investigate the safety and efficacy of DRA for CAG and PCI.

DETAILED DESCRIPTION:
Based on the results that radial approach (RA) reduced mortality and bleeding complications compared with femoral approach (FA), RA has become the standard of care for coronary angiography (CAG) and percutaneous coronary intervention (PCI). RA provides better comfortability for the patients and immediate mobilization after CAG or PCI. Therefore, 2018 ESC/EACTS guidelines recommend RA as the standard approach, unless there are overriding procedural considerations.

Operators usually prefer right RA because most of the operators are right-handed and right hand of the patient is closer to the operator. In contrast, longer distance to the left radial artery cause neck or back sprain of the operators, especially when the height of the operator is short, or the patient is obese. Nevertheless, left RA might be easier to manipulate catheter because of less tortuosity compared to the right RA and similar approach curvature with FA. Left RA also gives a chance to the right-handed patients to use their right hand freely.

Recently, the left distal radial approach (DRA) has been introduced as a feasible and safe alternative route of the radial artery. The left hand in the prone position is placed either on the left groin or beside the left hip according to operator preference. The operator punctures the distal radial artery around the anatomical snuffbox. After the first report for the feasibility and safety of left DRA in 70 patients, Lee et al. demonstrated that the success rates of arterial puncture, CAG and PCI were 95.5% (191/200), 100% (187/187), and 98.9% (86/87), respectively. The complication rates were only 7.9% including 14 (7.4%) minor hematomas and one (0.5%) arterial dissection. No serious complications were occurred such as distal radial artery occlusion, perforation, pseudoaneurysm, or arteriovenous fistula. Several studies for DRA also showed similar favorable results regarding procedural success and bleeding complications.

Radial arterial occlusion after RA remains an unsolved problem. According to the Leipzig prospective vascular ultrasound registry, the occlusion rate of radial artery was 14.4% in case of 5Fr sheath and 33.1% in 6Fr sheath, respectively. In this point of view, DRA could be a promising solution to lower the incidence rate of arterial occlusion. Moreover, DRA can have a potential benefit in patients requiring arteriovenous fistula and in patients who need the radial artery as a conduit for coronary artery bypass graft because of the absence of radial injury.

There is still lack of evidence for DRA regarding the feasibility, safety, effective time for hemostasis and hemostasis method. Unknown complications related to DRA also should be addressed. Therefore, this prospective multicenter registry aimed to investigate the safety and efficacy of DRA for CAG and PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years who planned coronary angiography
* Patients with palpable distal radial artery
* Patients who give informed consent

Exclusion Criteria:

* Patients with small or non-palpable distal radial artery
* Positive result in modified Allen test (suspicious of single blood supply)
* Pregnant women, possible candidate for pregnancy, or breastfeeding women
* Patients who are deemed unsuitable by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need coronary angiography will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
Success rate of coronary angiography | Through procedure completion, up to 6 hours
  Success rate of coronary angiography (%)
Success rate of percutaneous coronary intervention | Through procedure completion, up to 6 hours
  Success rate of percutaneous coronary intervention (%)

SECONDARY OUTCOMES:
Success rate of distal radial artery puncture | Through procedure completion, up to 6 hours
  Success rate of distal radial artery puncture (%)
Puncture time | Through procedure completion, up to 6 hours
  Puncture time (minute)
Hemostasis time | Through procedure completion, up to 24 hours
  Hemostasis time (minute)
Puncture-related complications | Up to 1 month
  Puncture-related complications (%)
Total procedure time | Through procedure completion, up to 6 hours
  Total procedure time (minutes)
Total fluoroscopic time | Through procedure completion, up to 6 hours
  Total fluoroscopic time (minute)
Total fluoroscopic dose | Through procedure completion, up to 6 hours
  Total fluoroscopic dose (Gray/cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital
Locations (14):
- South Korea (14):
  - Yongin Severance Hospital, Yongin-si, Kyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin Univeristy Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - GangNeung Asan Hospital, Gangneung
  - Inje University Ilsan Paik Hospital, Goyang
  - Dongguk University Gyeongju Hospital, Gyeongju
  - Uvis Hospital, Incheon
  - The Catholic university of Korea Uijeongbu St. Mary's hospital, Uijeongbu-si
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roh JW, Heo SJ, Lee OH, Im E, Cho DK, Lee JW, Lee BK, Yoo SY, Lee SY, Kim CJ, Jin HY, Park JS, Heo JH, Kim DH, Lee JB, Kim DK, Bae JH, Lee SY, Lee SH, Kim Y. Distal Radial Access and Women: Implications for Access Site Outcomes in Coronary Procedures. J Am Heart Assoc. 2025 Apr 15;14(8):e036285. doi: 10.1161/JAHA.124.036285. Epub 2025 Apr 10. PMID 40207479
- [Derived] Jin IT, Roh JW, Lee OH, Im E, Cho DK, Lee JW, Lee BK, Yoo SY, Lee SY, Kim CJ, Jin HY, Park JS, Heo JH, Kim DH, Lee JB, Kim DK, Bae JH, Lee SY, Lee SH, Kim Y. Feasibility of Distal Radial Access in High Bleeding Risk Patients Who Underwent Percutaneous Coronary Intervention. Korean Circ J. 2025 Apr;55(4):291-301. doi: 10.4070/kcj.2024.0239. Epub 2024 Nov 14. PMID 39733460
- [Derived] Lee JW, Kim Y, Lee BK, Yoo SY, Lee SY, Kim CJ, Jin HY, Park JS, Heo JH, Kim DH, Lee JB, Kim DK, Bae JH, Lee SY, Lee SH. Distal Radial Access for Coronary Procedures in a Large Prospective Multicenter Registry: The KODRA Trial. JACC Cardiovasc Interv. 2024 Feb 12;17(3):329-340. doi: 10.1016/j.jcin.2023.11.021. PMID 38355261